CLINICAL TRIAL: NCT00719238
Title: A Pilot Study to Promote Maternal and Infant Oral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Connecticut Health Foundation (Other)
Responsible Party: Susan Reisine, University of Connecticut School of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07-093-02; CTF2007
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2008-07-21 (Estimated); Status verified 2008-07

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Nutritional Status; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Nutrition plus education
- 2 (Active Comparator)
  Interventions: Behavioral: Education only

INTERVENTIONS:
Behavioral: Nutrition plus education — Nutritional instruction in small groups plus education
  Arms: 1
Behavioral: Education only — Educational video and pamphlets
  Arms: 2

SUMMARY:
The long term goals of this project are to develop and implement a combined prenatal and postnatal intervention to decrease early childhood caries. The program is based on risk assessment, diet intervention and counseling. To accomplish these goals a pilot study is needed to determine: 1) The ability to recruit and retain pregnant mothers in an intervention program; 2) The levels of S. mutans in pregnant mothers; 3) The ability of a diet intervention to decrease S. mutans in pregnant mothers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over;
* Pregnant
* High S. mutans levels

Exclusion Criteria:

* Younger than 18;
* Other health conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Sugar intake | 3 months post partum

SECONDARY OUTCOMES:
mutans streptococci levels | 3 months post partum

CONTACTS AND LOCATIONS:
Overall Officials: Susan Reisine, PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States